CLINICAL TRIAL: NCT04086381
Title: Creatine Monohydrate Supplementation in Young, Healthy Vegetarian Adults and Its Effect on Brown Adipose Tissue Activation
Brief Title: Creatine Effect on Brown Adipose Tissue Activation
Acronym: CreaBAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University (Other)
Responsible Party: Principal Investigator, Patrick Schrauwen, Principal Investigator, Maastricht University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NL64709.068.18
Record Dates: First submitted 2019-09-10; First posted 2019-09-11 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Diet-induced Thermogenesis; Brown Adipose Tissue Activation
Keywords: Brown adipose tissue; Creatine monohydrate; Diet-induced thermogenesis
MeSH Terms: interventions — Creatine

STUDY DESIGN:
Intervention Model Description: A double-blind, randomised, controlled, cross-over intervention trial.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Oral injestion of 20 grams of creatine monohydrate daily
  Interventions: Dietary Supplement: Creatine monohydrate
- Placebo (Placebo Comparator): Oral injestion of 20 grams of cellulose daily
  Interventions: Dietary Supplement: placebo cellulose

INTERVENTIONS:
Dietary Supplement: Creatine monohydrate — 5 grams of creatine monohydrate, four times daily, for 9 consecutive days.
  Arms: Intervention
Dietary Supplement: placebo cellulose — oral ingestion of placebo containing 20 gram cellulose daily
  Arms: Placebo

SUMMARY:
Pre-clinical studies indicate that creatine may play a substantial role in diet-induced thermogenesis and may have a profound effect on energy balance. A recent retrospective study of BAT activation on PET-CT scans in humans showed a positive association with the estimated renal creatinine clearance and BAT activation, possibly linking creatine metabolism in humans to BAT activity. In humans, so far little options are available to activate brown adipose tissue. The most potent intervention to activate BAT is via cold, which has previously been shown to have metabolic effects in humans. Provided the potential health benefits of brown adipose tissue activation in humans, and provided the role of brown fat in diet induced thermogenesis, we here aim to determine whether creatine monohydrate supplementation can increase diet-induced thermogenesis and activate brown adipose tissue in humans.

ELIGIBILITY:
Inclusion Criteria:

* Male or female;
* 18 to 30 years of age;
* Consuming a vegetarian diet;
* BMI 20-25 kg/m2.

Exclusion Criteria:

* Not meeting all inclusion criteria;
* Non-vegetarian diet;
* Excessive alcohol and/or drug abuse;
* Significant allergies or intolerances concerning the study products;
* Participation in another biomedical study within 1 month before the first study visit, possibly interfering with the study results;
* Medication use known to hamper subject's safety during the study procedures;
* Subjects with contra-indications for MRI and/or PET-CT;
* Subjects who do not want to be informed about unexpected medical findings;
* Subjects who do not want that their treating physician to be informed;
* Co-morbidities to which the intervention or program that may pose as a complicating factor;
* Inability to participate and/or complete the required measurements;
* PET-CT scan in the last 12 months.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-01-22 (Actual)

PRIMARY OUTCOMES:
Brown adipose tissue activation through 18F-FDG PET-MRI | Day 10 of protocol
  Standard Uptake Value (SUV)

SECONDARY OUTCOMES:
Diet-induced thermogenesis through indirect calorimetry | Day 8 of protocol
  Whole body energy expenditure in kJ/kg/min
Posphocreatine (PCr) Recovery through 31P-MRS | Day 9 of protocol
  Halftime of PCr Recovery

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Connell NJ, Doligkeit D, Andriessen C, Kornips-Moonen E, Bruls YMH, Schrauwen-Hinderling VB, van de Weijer T, van Marken-Lichtenbelt WD, Havekes B, Kazak L, Spiegelman BM, Hoeks J, Schrauwen P. No evidence for brown adipose tissue activation after creatine supplementation in adult vegetarians. Nat Metab. 2021 Jan;3(1):107-117. doi: 10.1038/s42255-020-00332-0. Epub 2021 Jan 18. PMID 33462512